CLINICAL TRIAL: NCT05477316
Title: A Single-arm Pilot Study, to Assess the Efficacy of Cerebellar IMRT Combined With Cerebral SRS in Patients With Brain Metastases That Are Predominantly in the Posterior Fossa - a Novel Treatment Approach
Brief Title: A Study to Assess the Efficacy of Cerebellar IMRT Combined With Cerebral SRS in Patients With Brain Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Meirrovitz Amichay, Principle investigator, oncologist and radiation specialist, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0930-20
Record Dates: First submitted 2021-12-12; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Brain Metastases; Posterior Fossa Lesion; Cerebral Lesion
Keywords: Brain Metastases; Posterior Fossa; Cerebellum; Cerebral Lesion; Cerebrum
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Intensity-modulated Radiation Therapy (IMRT)/VMAT with integrated boost to the cerebellum and metastases and Stereotactic Radiosurgery (SRS) to the cerebral metastases as a novel treatment combination for brain metastases
  Interventions: Radiation: Radiation treatment

INTERVENTIONS:
Radiation: Radiation treatment — Radiation treatment of IMRT to the cerebellum and SRS to the cerebrum

SUMMARY:
A single-arm pilot study, to assess the efficacy of cerebellar IMRT combined with cerebral SRS in patients with brain metastases that are predominantly in the posterior fossa - a novel treatment approach

DETAILED DESCRIPTION:
This study includes patients with brain metastases, presenting with more than 5 cerebellar lesions and less than 10 cerebral lesions. This is a pilot study assessing the efficacy of a novel, combined treatment approach involving Intensity-modulated Radiation Therapy (IMRT)/ Volumetric Modulated Arc Therapy (VMAT), with or without integrated boost to metastases, administered to the posterior fossa, and Stereotactic Radiosurgery (SRS) administered to cerebral lesions. This is opposed to the current recommended treatment approach for such cases, being whole brain radiotherapy (WBRT). While an effective treatment with respect to lesion control, WBRT is not ideal as the total deliverable dose is limited to 30 Gy due to toxicity. In addition, this technique is responsible for major side effects, especially neurocognitive deterioration.

There are select cases of multiple brain metastases which are predominantly found in the posterior fossa. Rectal cancer is one such notorious example, however this type of spread is not limited to one region.

The investigators hypothesize that utilizing the novel combinational treatment approach of IMRT and SRS in cerebral and cerebellar brain metastases will improve long term brain control, maintain the patients' cognitive function and potentially improve overall survival, as the need for potent WBRT will become obsolete.

Patients with multiple brain metastases present in the cerebrum and cerebellum will be treated with SRS and IMRT respectively, simultaneously (within 3 weeks of one another). Brain MRI scans will be performed before commencement of the novel treatment approach, at two month after RT, and then every 3 months, or as indicated clinically, after treatment start. Concurrently at each MRI scan time point, patients will be assessed based on brain and whole-body metastatic progression by RECIST. Patients will also be assessed for central nervous system (CNS) - progression free survival (PFS) and body-PFS, cognitive function, quality of life and overall survival status via standardized follow-up tests.

ELIGIBILITY:
Inclusion criteria

1. Presence of multiple brain metastasis, predominantly in the posterior fossa: more than 5 metastases in the cerebellum, and less than 10 metastases in the cerebrum, visible on MRI, regardless of tumor origin.
2. Provided written informed consent.
3. Be male or female and at least 18 years of age on the day of signing informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. A minimum life expectancy of at least 3 months
6. Female patients:

   1. Willing to use adequate contraceptive measures until 6 weeks after the final dose of study treatment
   2. Not breast feeding
   3. Have a negative pregnancy test prior to the start of dosing if of childbearing potential or have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:
   4. i. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments ii. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution iii. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
7. Male patients who are willing to use barrier contraception (i.e. condoms) until 4 months after the final dose of study treatment.

Exclusion criteria

1. Prior treatment with Whole brain radiation (WBRT) (previous SRS is allowed for limited, up to 4 metastases, six month or more prior to the study treatment, and the index metastases should be all new)
2. An investigational drug within five half-lives of the compound.
3. Spinal cord compression unless asymptomatic and stable.
4. Leptomeningeal disease.
5. Moderate or severe symptomatic brain metastases defined as per Radiation therapy Oncology Group acute morbidity grade 3 to 4.

   Note: Grade 3 refers to neurological findings requiring hospitalization for initial management. Grade 4 refers to serious neurological impairment including paralysis, coma or seizures more than three times per week despite medication and requires hospitalization.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Involvement in the planning and conduct of the study
8. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain control: Central Nervous System (CNS)- Progression Free Survival (PFS) | Change in lesion size in the whole body will be followed and assessed at screen, 2 month after radiation treatment, then every 3 month until the date of first documented progression or date of death from any cause, up to 10 years.
  Metastatic brain lesions treated with IMRT/SRS will be tracked and measured using MRI. Disease in the brain and systemically will be assessed by RECIST.

SECONDARY OUTCOMES:
Cognitive function | Change in patient cognitive function will be followed and assessed at screen, 2 month after radiation treatment, then every 3 month, until the date of first documented progression or date of death from any cause, up to 10 years.
  Patient cognitive function will improve after study treatment (Hopkines verbal learning test (HVLT), Trail Making Test (TMT) A + B, Controlled Oral Word Association Test (COWAT) and clock drawing test). Cognitive functions will be univariately compared between the groups using the Student's t-test or the Mann-Whitney Ranks test. We will also perform multivariate analyses using either linear regression of Poisson regression, depending on the outcomes distribution.
Quality of life (QOL) | Change in patient QOL will be followed and assessed at screen, 2 month after radiation treatment, then every 3 month, until the date of first documented progression or date of death from any cause, up to 10 years.
  Patient QOL will improve after study treatment. QOL will be evaluated due to score in four questionnaires: European Organisation for. Research and Treatment of Cancer (EORTC) QLQ C30, The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT), The Pittsburgh Sleep Quality Index (PSQI) and Hospital Anxiety and Depression Scale (HADS). Cognitive functions will be univariately compared between the groups using the Student's t-test or the Mann-Whitney Ranks test. We will also perform multivariate analyses using either linear regression of Poisson regression, depending on the outcomes distribution.
Overall survival (OS) | Status will be checked at every visit and follow up, until the date of death from any cause, up to 10 years.
  Patient OS will be assessed via timely patient follow-ups on survival status

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutt R, Dawson G, Cheuk AV, Fosmire H, Moghanaki D, Kelly M, Jolly S. Palliative Radiotherapy for the Management of Metastatic Cancer: Bone Metastases, Spinal Cord Compression, and Brain Metastases. Fed Pract. 2015 May;32(Suppl 4):12S-16S. PMID 30766118
- [Background] Nayak L, Lee EQ, Wen PY. Epidemiology of brain metastases. Curr Oncol Rep. 2012 Feb;14(1):48-54. doi: 10.1007/s11912-011-0203-y. PMID 22012633
- [Background] Achrol AS, Rennert RC, Anders C, Soffietti R, Ahluwalia MS, Nayak L, Peters S, Arvold ND, Harsh GR, Steeg PS, Chang SD. Brain metastases. Nat Rev Dis Primers. 2019 Jan 17;5(1):5. doi: 10.1038/s41572-018-0055-y. PMID 30655533
- [Background] Martinez P, Mak RH, Oxnard GR. Targeted Therapy as an Alternative to Whole-Brain Radiotherapy in EGFR-Mutant or ALK-Positive Non-Small-Cell Lung Cancer With Brain Metastases. JAMA Oncol. 2017 Sep 1;3(9):1274-1275. doi: 10.1001/jamaoncol.2017.1047. PMID 28520828
- [Background] Godfrey SE. Estrogen receptors. Am J Clin Pathol. 1989 May;91(5):629-30. doi: 10.1093/ajcp/91.5.629. No abstract available. PMID 2718965
- [Background] Greene-Schloesser D, Robbins ME, Peiffer AM, Shaw EG, Wheeler KT, Chan MD. Radiation-induced brain injury: A review. Front Oncol. 2012 Jul 19;2:73. doi: 10.3389/fonc.2012.00073. eCollection 2012. PMID 22833841
- [Background] Tsao MN, Xu W, Wong RK, Lloyd N, Laperriere N, Sahgal A, Rakovitch E, Chow E. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2018 Jan 25;1(1):CD003869. doi: 10.1002/14651858.CD003869.pub4. PMID 29365347
- [Background] Soike MH, Hughes RT, Farris M, McTyre ER, Cramer CK, Bourland JD, Chan MD. Does Stereotactic Radiosurgery Have a Role in the Management of Patients Presenting With 4 or More Brain Metastases? Neurosurgery. 2019 Mar 1;84(3):558-566. doi: 10.1093/neuros/nyy216. PMID 29860451
- [Background] Sahgal A, Aoyama H, Kocher M, Neupane B, Collette S, Tago M, Shaw P, Beyene J, Chang EL. Phase 3 trials of stereotactic radiosurgery with or without whole-brain radiation therapy for 1 to 4 brain metastases: individual patient data meta-analysis. Int J Radiat Oncol Biol Phys. 2015 Mar 15;91(4):710-7. doi: 10.1016/j.ijrobp.2014.10.024. PMID 25752382
- [Background] Sahgal A, Ruschin M, Ma L, Verbakel W, Larson D, Brown PD. Stereotactic radiosurgery alone for multiple brain metastases? A review of clinical and technical issues. Neuro Oncol. 2017 Apr 1;19(suppl_2):ii2-ii15. doi: 10.1093/neuonc/nox001. PMID 28380635
- [Background] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- [Background] Nabors LB, Ammirati M, Bierman PJ, Brem H, Butowski N, Chamberlain MC, DeAngelis LM, Fenstermaker RA, Friedman A, Gilbert MR, Hesser D, Holdhoff M, Junck L, Lawson R, Loeffler JS, Maor MH, Moots PL, Morrison T, Mrugala MM, Newton HB, Portnow J, Raizer JJ, Recht L, Shrieve DC, Sills AK Jr, Tran D, Tran N, Vrionis FD, Wen PY, McMillian N, Ho M; National Comprehensive Cancer Network. Central nervous system cancers. J Natl Compr Canc Netw. 2013 Sep 1;11(9):1114-51. doi: 10.6004/jnccn.2013.0132. PMID 24029126
- [Background] Sahgal A. Point/Counterpoint: Stereotactic radiosurgery without whole-brain radiation for patients with a limited number of brain metastases: the current standard of care? Neuro Oncol. 2015 Jul;17(7):916-8. doi: 10.1093/neuonc/nov087. No abstract available. PMID 26092877
- [Background] Sahgal A, Larson D, Knisely J. Stereotactic radiosurgery alone for brain metastases. Lancet Oncol. 2015 Mar;16(3):249-50. doi: 10.1016/S1470-2045(14)71106-4. No abstract available. PMID 25752547
- [Background] Mohammadi AM, Recinos PF, Barnett GH, Weil RJ, Vogelbaum MA, Chao ST, Suh JH, Marko NF, Elson P, Neyman G, Angelov L. Role of Gamma Knife surgery in patients with 5 or more brain metastases. J Neurosurg. 2012 Dec;117 Suppl:5-12. doi: 10.3171/2012.8.GKS12983. PMID 23205782
- [Background] Grandhi R, Kondziolka D, Panczykowski D, Monaco EA 3rd, Kano H, Niranjan A, Flickinger JC, Lunsford LD. Stereotactic radiosurgery using the Leksell Gamma Knife Perfexion unit in the management of patients with 10 or more brain metastases. J Neurosurg. 2012 Aug;117(2):237-45. doi: 10.3171/2012.4.JNS11870. Epub 2012 May 25. PMID 22631694
- [Background] Rava P, Leonard K, Sioshansi S, Curran B, Wazer DE, Cosgrove GR, Noren G, Hepel JT. Survival among patients with 10 or more brain metastases treated with stereotactic radiosurgery. J Neurosurg. 2013 Aug;119(2):457-62. doi: 10.3171/2013.4.JNS121751. Epub 2013 May 10. PMID 23662828
- [Background] Chang WS, Kim HY, Chang JW, Park YG, Chang JH. Analysis of radiosurgical results in patients with brain metastases according to the number of brain lesions: is stereotactic radiosurgery effective for multiple brain metastases? J Neurosurg. 2010 Dec;113 Suppl:73-8. doi: 10.3171/2010.8.GKS10994. PMID 21121789
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Gerstenecker A, Nabors LB, Meneses K, Fiveash JB, Marson DC, Cutter G, Martin RC, Meyers CA, Triebel KL. Cognition in patients with newly diagnosed brain metastasis: profiles and implications. J Neurooncol. 2014 Oct;120(1):179-85. doi: 10.1007/s11060-014-1543-x. Epub 2014 Jul 18. PMID 25035099
- [Background] Trifiletti DM, Lee CC, Winardi W, Patel NV, Yen CP, Larner JM, Sheehan JP. Brainstem metastases treated with stereotactic radiosurgery: safety, efficacy, and dose response. J Neurooncol. 2015 Nov;125(2):385-92. doi: 10.1007/s11060-015-1927-6. Epub 2015 Sep 4. PMID 26341374
- See also: Related Info — http://www.choosingwisely.org/astro-releases-second-list/
- See also: Related Info — https://www.researchgate.net/publication/346391013_Stereotactic_Radiosurgery_versus_Whole-brain_Radiation_Therapy_for_Patients_with_4-15_Brain_Metastases_A_Phase_III_Randomized_Controlled_Trial